CLINICAL TRIAL: NCT06468683
Title: A Phase I Clinical Study to Evaluate the Safety, Pharmacokinetics, and Preliminary Efficacy of F01 in Patients With Moderate-to-severe Refractory Systemic Lupus Erythematosus
Brief Title: F01 in the Treatment of Moderate-to-severe Refractory Systemic Lupus Erythematosus
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Simnova Biotechnology Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNC 103-CD19CAR NK-104
Record Dates: First submitted 2024-05-31; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-05

CONDITIONS: Lupus Erythematosis
Keywords: Moderate-to-severe refractory systemic lupus erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: After preconditioning with chemotherapy, F01 will be evaluated. (Experimental): Assigned Interventions
  Interventions: Biological: After preconditioning with chemotherapy, F01 will be evaluated.

INTERVENTIONS:
Biological: After preconditioning with chemotherapy, F01 will be evaluated. — Biological: 0.5-3×10^9 CAR+NK Cells, Treatment follows a lymphodepletion Drug: Fludarabine: 25-30 mg/m^2 (D-5~D-3) Drug: Cyclophosphamide: 250-300 mg/ m^2 (D-5~D-3)

SUMMARY:
This is a phase I clinical study to evaluate the safety , pharmacokinetic profile, and preliminary efficacy of F01 in patients with moderate-to-severe refractory systemic lupus erythematosus.

DETAILED DESCRIPTION:
Approximately up to about 50 participants with moderate-to-severe refractory systemic lupus erythematosus are planned to enroll. This study is divided into two stages: dose escalation and dose extension.

ELIGIBILITY:
Inclusion Criteria:

- Participants must meet all of the following inclusion criteria to be enrolled in the study:

1. Age ≥18 and ≤65 years old, gender unlimited.
2. Subjects with moderate-to-severe refractory SLE must meet all of the following criteria:

   * Diagnosis of SLE at least 24 weeks prior to screening in accordance with the European Federation of Rheumatological Societies (EULAR)/American College of Rheumatology (ACR) 2019 SLE classification criteria at screening;
   * Applicants must meet one of the following criteria at screening: a. positive for antinuclear antibody (ANA); b. Positive anti-dsDNA antibody;c. Positive anti-Smith antibody;
   * SLEDAI-2000 score ≥ 8 at screening
3. Have received adequate standard doses of glucocorticoids, antimalarials, immunosuppressants/immunomodulators, and at least one biologic agent for at least 2 months prior to screening, with a stable dose > disease remaining active after 2 weeks of treatment. Oral glucocorticoids must meet the following requirements: 1) Prednisone (or equivalent) ≥ 7.5 mg/day and ≤ 60 mg/day. 2) When used in combination with immunosuppressants and/or biologics, there is no minimum daily dose requirement for glucocorticoids. The blood routine within 7 days of clear drenching conditioning chemotherapy meets the following requirements:

   * Absolute neutrophil value (ANC) ≥ 1.5×109/L;
   * Hemoglobin (Hb) ≥ 80g/L;
   * Platelet count (PLT) ≥ 50×109/L.
4. Adequate hepatic, renal, lung, and cardiac function, defined as:

   1. Serum ALT and AST ≤ 2.5 times the upper limit of normal;
   2. Total bilirubin ≤ 1.5 times the upper limit of normal, except for patients with Gilbert's syndrome, where total bilirubin must be ≤ 3.0 times the upper limit of normal;
   3. creatinine clearance (estimated by Cockcroft Gault's formula) (Appendix 1) ≥ 50 ml/min;
   4. Oxygen saturation of ≥ 92% in non-oxygenated conditions under indoor ventilation; No clinically significant pleural effusion;
   5. Left ventricular ejection fraction ≥ 50%; Echocardiography to confirm the absence of pericardial effusion; There were no clinically significant abnormal findings on ECG.
5. Subjects receiving hematopoietic growth factor supportive therapy, including erythropoietin (EPO), granulocyte colony-stimulating factor (G-CSF), granulocyte macrophage-colony-stimulating factor (GM-CSF) and platelet agonists (TPO), etc., must have a 2-week gap between the last growth factor supportive therapy and the screening period evaluation; Patients receiving blood product transfusions should have at least 1 week between the screening platelet assessment and the last platelet transfusion, and at least 2 weeks between the screening hemoglobin assessment and the last red blood cell transfusion.
6. During the screening period, female subjects of childbearing potential must have a negative serum pregnancy test result (women who have been surgically sterilized or postmenopausal for at least 2 years are considered not of childbearing potential). Female subjects of childbearing potential and male subjects must use a highly effective method of contraception throughout the clinical study period and for 1 year after the last dose of study treatment; At the same time, a commitment should be made not to donate eggs (oocytes, oocytes)/sperm for assisted reproduction within 1 year after the last study treatment.
7. Voluntarily participate in clinical trials and sign informed consent.

Exclusion Criteria:

* Subjects who meet any of the following exclusion criteria will not be admitted to this clinical study:

  1. Known allergies, hypersensitivity, intolerance, or contraindications to F01 or any ingredient of drugs that may be used in the study (including fludarabine, cyclophosphamide, tocilizumab), or subjects who have had severe allergic reactions in the past.
  2. Severe lupus nephritis (defined as urine protein >6g/24 hours or serum creatinine >2.5mg/dL or 221μmol/L) within 3 months prior to screening, or requiring active nephritis with drugs prohibited by the protocol, or requiring hemodialysis or treatment with prednisone ≥100mg/d or equivalent glucocorticoids ≥for 14 days.
  3. Previous history or pathological changes of clinically significant central nervous system disease, including but not limited to lupus encephalopathy, seizures, cerebrovascular accident (ischemia/hemorrhage), dementia, cerebellar disease, organic encephalopathy syndrome, encephalitis, central nervous system vasculitis, or psychiatric disease.
  4. Combined with severe pulmonary diseases, such as pulmonary hypertension with World Health Organization functional classification ≥ level 3, requiring oxygen therapy with an oxygen storage mask or non-invasive or invasive ventilator to assist breathing at screening;
  5. Unstable cardiovascular function:

     1. Myocardial infarction within 6 months prior to screening;
     2. Unstable angina within 3 months prior to screening;
     3. Uncontrolled, clinically significant cardiac arrhythmias (e.g., sustained ventricular tachycardia, ventricular fibrillation, torsades de pointes);
     4. Mobitz type II. second-degree or third-degree atrioventricular block;
     5. New York Cardiac Function Association Class ≥ 3 congestive heart failure;
     6. Poorly controlled hypertension (systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 100 mmHg) or concomitant hypertensive crisis or hypertensive encephalopathy;
  6. Patients with a history of concomitant malignancy, including tumor-associated polymyositis/dermatomyositis. Patients with non-melanoma skin cancer, carcinoma in situ of the cervix, local prostate cancer, low-stage bladder cancer, ductal carcinoma in situ, or patients who have no evidence of recurrence in the past 2 years and do not need treatment are excluded.
  7. Uncontrolled active bacterial, viral, fungal, mycobacterial infection or other infections requiring treatment with intravenous antibiotics, antiviral or antifungal drugs within 14 days prior to drenching conditioning chemotherapy; However, these drugs can be used for prophylactic treatment (including intravenous use).
  8. Risk of active tuberculosis at screening, regardless of completion of adequate treatment, including the presence of signs or symptoms of active tuberculosis (such as fever, cough, night sweats, and weight loss) as judged by the investigator at screening; Chest imaging (e.g., chest x-ray, chest CT scan) documented at screening or at any time within 6 months prior to screening showing active tuberculosis; Evidence of latent tuberculosis infection, such as a positive γ-interferon release test, at screening.
  9. Active hepatitis B virus (HBV), hepatitis C virus (HCV) infection at screening. Subjects who are HBsAg positive and/or HBcAb positive but HBV-DNA negative, and/or HCVAb positive but HCV-RNA negative are allowed to be enrolled (if the site report includes a range of reference values, the upper limit of normal for HBV-DNA and HCV-RNA tests is based on the test values of each site, and higher than the upper limit of test values is defined as "positive"; If the site report only shows "negative/positive", the positive is based on the test report result).
  10. Known serum HIV virus antibody positivity or history of active HIV infection, as well as syphilis antibody positive.
  11. Received the following treatments within the prescribed time frame prior to drenching conditioning chemotherapy:

      1. Received autologous/allogeneic hematopoietic stem cell transplantation within 3 months;
      2. Received ultraviolet radiation therapy within 6 weeks;
      3. Received macromolecule therapy (excluding anti-CD20 monoclonal antibodies) within 4 weeks or 3 half-lives (whichever is longer); Received anti-CD20 monoclonal antibody therapy within 4 weeks;
      4. Received small molecule targeted therapy within 2 weeks or 3 half-lives (whichever is longer);
      5. Major surgery or live vaccination within 4 weeks;
      6. Received a trial treatment within 4 weeks (except in the definitive placebo control group);
  12. Pregnant or lactating women.
  13. Use of concomitant medications/concomitant treatments expressly prohibited by the protocol during the screening period.
  14. Presence of any life-threatening disease, medical condition, or organ system dysfunction that, in the opinion of the investigator, may affect the subject's safety or study compliance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measures | 12 weeks
  The proportion of subjects with AEs and SAEs
Primary Outcome Measures | 4 weeks
  The proportion of subjects with DLT

SECONDARY OUTCOMES:
Secondary Outcome Measures | 48 weeks
  Efficacy of F01 cells in moderate-to-severe refractory systemic lupus erythematosus
Secondary Outcome Measures | 96 weeks
  Cellular kinetics [ Time Frame: 96 weeks] The maximum concentration (Cmax)
Secondary Outcome Measures | 96 weeks
  Cellular kinetics [ Time Frame: 96 weeks] the time to reach the highest concentration (Tmax)
Secondary Outcome Measures | 96 weeks
  Cellular kinetics [ Time Frame: 96 weeks] the area under the curve of the drug time (AUC0-last)
Secondary Outcome Measures | 96 weeks
  Cellular kinetics [ Time Frame: 96 weeks] the last detectable concentration point (Clast)
Secondary Outcome Measures | 96 weeks
  Cellular kinetics [ Time Frame: 96 weeks] the time of the last detectable concentration (Tlast), etc.
Secondary Outcome Measures | 96 weeks
  Cellular kinetics [ Time Frame: 96 weeks] dynamic changes in cytokine levels in the subject's peripheral blood at baseline and after dosing; The number of cases, positive rate
Secondary Outcome Measures | 96 weeks
  Cellular kinetics [ Time Frame: 96 weeks] duration of anti-CAR and IL-15 antibodies (ADA)

OTHER OUTCOMES:
Exploratory | 96 weeks
  Explore the correlation between the concentration of PK and PD and efficacy and safety by CTCAE v5.0
Exploratory | 96 weeks
  Explore the correlation between KIR mismatch and efficacy and safety by CTCAE v5.0
Exploratory | 96 weeks
  Immunogenicity study of Cas9

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai jiaotong University School of Medicine,Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided